CLINICAL TRIAL: NCT02626039
Title: Characterization and Comparison of Drugable Mutations in Primary Tumors, Metastatic Tissue, Circulating Tumor Cells and Cell-Free Circulating DNA in Metastatic Breast Cancer Patients
Brief Title: Characterization & Comparison of Drugable Mutations in Primary and Metastatic Tumors, CTCs and cfDNA in MBCpatients
Acronym: MIRROR
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Other Study IDs: GOMHGUGM092013
Record Dates: First submitted 2015-10-15; First posted 2015-12-10 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; CTCs; cfDNA; genomics; somatic mutations
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Primary and Metastatic tumoral tissue (FFPE samples) and Blood samples

SUMMARY:
Characterization of the driver mutations in an individual metastatic breast cancer patient is critical for many reasons. Effective targeted therapies require identifying genomic alterations in the tumoral tissue. The scarce efficacy of many currently available targeted drugs may be due to the outbreak of resistant clones with different genotype that already present at the initiation of therapy. It is well known the intra-tumor heterogeneity with genetic and non-genetic factors considered as the origin of the tumor cell-clon composition. The acquisition of multiple mutations (driver and passenger), altogether with the stage of differentiation, according to the cancer stem cell hypothesis, confers to the tumor cells clinically important properties, such as resistance to therapies and seeding abilities.

Moreover, there is a current challenge in establishing whether the metastatic cells arise from the most aggressive and dominant clone in the primary tumor or the metastasic tissue diverges with substantial genetic changes very early in the evolution of the disease. Primary and metastatic tumor may have a close clonal relationship or evolve in parallel and acquire different genomic alterations. In the real life, it is plausible that both models coexist with different predominance according to the tumoral tissue and etiology.

The study hypothesizes that breast cancer metastases and primary tumors could harbor different genomic profiles related to genomic regions of interest in a clinically relevant proportion of metastatic breast cancer patients.

Moreover, the genomic aberrations found in the metastatic breast cancer tissue could also be detected in CTCs and circulating free DNA.

If true, CTCs and circulating free DNA would be convenient, non-invasive, easily accessible sources of genomic material for the analysis of mutations and other genomic aberrations.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer confirmed by radiologic findings
* ≥ 18 years old
* Able to give signed consent
* Availability to get the paraffin block of her primary tumor.
* First metastatic relapse or tumor regrowth while on treatment for metastatic disease (progressive disease while on treatment)
* Biopsy of the metastatic site clinically indicated

Exclusion Criteria:

* Inability to get a core sample from a metastatic site
* Bone disease only (the decalcification process usually prevents an appropriate genomic study).
* Unable to drawn peripheral blood
* Unable to give the informed consent
* Coagulation disorders
* ECOG status 3-4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with metastatic breast cancer in which FFPE samples from the primary tumors are available and in whom a biopsy of the metastatic relapse is clinically indicated.
  Investigators will offer enrollment to consecutively seen women who meet the entry criteria. Target enrollment is 40 patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Cohen's kappa coefficient to measure the inter-rater agreement for mutations and other genomic findings (categorical items) between the metastatic tissue and the primary tumor tissue in Metastatic Breast Cancer patients. | 26 months

SECONDARY OUTCOMES:
Number of somatic genomic findings (found in the primary and metastatic tumor) in circulating tumoral cells (CTC) and circulating free DNA(cfDNA) obtained from peripheral blood (liquid biopsy). | 26 months
Description of the mutations in analyzed genes in the primary tumor and in CTC/cfDNA for each patient. | 26 months
  Note: circulating tumor cells couldn't be sequenced

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Martín, Ph, Study Chair — Hospital General Universitario Gregorio Marañon
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Derived] Gonzalez-Rivera M, Picornell AC, Alvarez EL, Martin M. A Cross-Sectional Comparison of Druggable Mutations in Primary Tumors, Metastatic Tissue, Circulating Tumor Cells, and Cell-Free Circulating DNA in Patients with Metastatic Breast Cancer: The MIRROR Study Protocol. JMIR Res Protoc. 2016 Aug 16;5(3):e167. doi: 10.2196/resprot.6024. PMID 27531554